CLINICAL TRIAL: NCT00803842
Title: Evaluation of Erlotinib Pharmacokinetics During Doxycycline Treatment for Erlotinib-induced Rash
Brief Title: Erlotinib Pharmacokinetics During Doxycycline Treatment for Erlotinib-induced Rash
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution and decided not to continue with the study.
Sponsor: Northwestern University (Other)
Responsible Party: Mario E. Lacouture, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEL-120407
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: erlotinib; rash; supportive care
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Exanthema | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: doxycycline — Doxycycline (the study drug) will be provided to all subjects as 100 mg tablets. They will be allocated enough doxycycline to last them until their next scheduled visit. The doxycycline tablets should be taken orally (only) at a dosage of 100 mg every 12 hours. Administration of adequate amounts of fluid along with capsule and tablet forms of drugs in the tetracycline class is recommended to wash down the drugs and reduce the risk of esophageal irritation and ulceration. The doxycycline tablets should not be taken with foods that contain calcium. The absorption of doxycycline is reduced when taking bismuth subsalicylate. Duration of study period if 14 days

SUMMARY:
A side effect occurring in a majority of patients taking erlotinib (Tarceva®) consists of a skin rash. Sometimes, symptoms associated with the rash necessitate erlotinib dose reduction or discontinuation. Some physicians have successfully treated the erlotinib-induced rash with doxycycline. At the same time, it has been observed that in patients who develop the erlotinib rash, the cancers respond better to erlotinib treatment. This research study is designed to determine how well doxycycline treats the erlotinib rash and whether doxycycline affects the blood levels of erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older.
* Subjects must have started Tarceva® therapy within three (3) days of trial enrollment.
* Patients must have signed informed consent prior to registration on study.
* Currently receiving erlotinib therapy at 150 mg per day for locally advanced or metastatic NSCLC.
* Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must utilize barrier methods in combination with spermicidal agents for contraception when engaging in sexual intercourse. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Exclusion Criteria:

* Allergy to tetracyclines.
* Use of concurrent agents for papulopustular rash.
* Currently receiving anticancer agents other than erlotinib.
* Inability to interrupt other antibiotic therapy.
* Current use of topical steroids
* Current use of systemic immunosuppressants (e.g., methotrexate, cyclosporine, azathioprine, mycophenolate mofetil)
* Photosensitivity or lupus erythematosus.
* Active gastroesophageal reflux disease.
* Women who have a positive pregnancy test or are lactating by history.
* ECOG performance status ≤3.
* Self report of current smoking or history of smoking within 60 days of screening, or positive urine cotinine test.
* Current use of agents that are known to be strong inducers or inhibitors of CYTP3A4:

  * inhibitors: atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfi navir, ritonavir, saquinavir, telithromycin, troleandomycin (TAO), voriconazole, grapefruit or grapefruit juice
  * inducers: rifampicin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, and St. John's Wort
* Impaired hepatic function (≤ 30 days before randomization):

  * Alkaline phosphatase > 3x ULN
  * Aspartate aminotransferase (AST) > x ULN
  * Alanine aminotransferase (ALT) > 3 x ULN
  * Total Bilirubin > 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether administration of doxycycline affects erlotinib PK | 14 days

SECONDARY OUTCOMES:
Secondarily, this study aims to investigate the relationship between erlotinib AUC and rash severity and to evaluate the efficacy of doxycycline in rash management. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lacouture, MD, Principal Investigator — Northwestern University